CLINICAL TRIAL: NCT00456573
Title: Local and Systemic Cytokine Profiles in Children With Obstructive Sleep Apnea and Controls
Brief Title: Cytokine Profiles in Children With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 002 (14437B)
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Pediatric Obstructive sleep apnea syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: tonsillectomy — medically indicated tonsillectomy in subjects with and without OAS

SUMMARY:
The purpose of this study is to compare the cytokine profile of tonsillar and peripheral blood mononuclear cells in patients with obstructive sleep apnea (OSA) and to compare the blood mononuclear cell cytokine secretion profile between patients with obstructive sleep apnea and controls without apnea.

DETAILED DESCRIPTION:
We will recruit subjects with OSA about to undergo adenotonsillectomy and collect a blood sample and portion of their tonsils after the induction of general anesthesia. The mononuclear cells will be isolated from both these tissues and stimulated with different markers and cytokines assayed and compared. We will also recruit patients with no symptoms of OSA undergoing unrelated elective surgery and ascertain the absence of OSA by having the parents fill out a sleep questionnaire. We will then collect blood samples from these patients after the induction of anesthesia and examine the cytokine secretion profile and compare it to that of the children with OSA.

ELIGIBILITY:
Inclusion Criteria:

* OSA documented by polysomnography and clinical symptoms.
* Patients with no symptoms of OSA and negative sleep questionnaire.

Exclusion Criteria:

* Significant systemic disease except mild asthma

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2008-09-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
levels of cytokines released from PBMCs of OAS subjects and controls | just prior to surgery

SECONDARY OUTCOMES:
cytokine level comparison between PBMCs and tonsillar lymphocytes within OAS groups | at time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fuad M Baroody, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States